CLINICAL TRIAL: NCT05887518
Title: The Effect of Sock Developed Wıth Wearable Technology for Patıents Undergoıng Transurethral Resectıon Surgery on the Development of Hypothermıa and Venous Thromboembolısm
Brief Title: The Effect of Sock Developed with Wearable Technology for TUR Surgery Patients on Hypothermia and Venous Thromboembolism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was canceled because the cost of the tests requested by the Turkish Medicines and Medical Devices Agency exceeded the project budget
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MU-BOZKUL-002
Record Dates: First submitted 2023-05-07; First posted 2023-06-02 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Transurethral Resection; Wearable Devices; Venous Thromboembolism; Hypothermia; Nurse
Keywords: transurethral resection; Wearable devices; venous thromboembolism; hypothermia; nurse
MeSH Terms: conditions — Venous Thromboembolism; Hypothermia | interventions — Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: Prospective, two-arm (1:1), randomised controlled, double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: A total of 70 patients in the sample group determined by randomisation will be divided according to the A and B groups formed by the same statistician in the computer environment. The information that the patients included in the research sample were assigned to group A and B according to the randomisation table will be kept by the consultant, and the socks with and without heating feature will be numbered from 1 to 70 according to the randomisation table and given to the practitioner so that the practitioner will be blinded when he/she does not know which sock has heating feature and which one does not. Thus, patients will be blinded as they do not know which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): In addition to the routine treatment and care practices of the operating theatre, the patients included in the study group will wear antiembolytic socks and warming socks to be developed with wearable technology. After the antiembolitic socks are put on the patients in the ward, the socks to be developed with wearable technology will be put on the study group before they are sent to the operating theatre and will be removed one day after the operation.
  The socks to be used in the research (heating socks developed with wearable technology will be developed by the researchers and patent application will be made.
  The application of socks to be developed with wearable technology in the research will be applied to all patients by the same executive. Verbal and written consent will be obtained from the patient/relative before the start of the study.
  Interventions: Device: Socks Developed with Wearable Technology
- CONTROL GROUP (No Intervention): In the control group, the same looking sock will be worn before the patient is sent to the operating theatre and will be removed one day after the operation.
  The sock to be used in the research will be developed by the researchers and a patent application will be made.
  Verbal and written consent will be obtained from the patient/relative before the start of the study. The data obtained from the patients will be recorded in the "Introductory Characteristics Form" and "Hypothermia Monitoring Form" before the TUR. The application of socks to be developed with wearable technology will be carried out in accordance with the following application steps.

INTERVENTIONS:
Device: Socks Developed with Wearable Technology — This new material will have the ability to prevent hypothermia by rewarming the patient when the body temperature drops below 360C and will reduce the risk of DVT that may develop in patients due to hypothermia. Thus, a single material will be used for two important complications of the surgical process, such as hypothermia and DVT, which negatively affect patient outcomes. This situation suggests that this material developed with an innovative approach will be more cost effective.
  Arms: EXPERIMENTAL GROUP

SUMMARY:
The aim of this study is to examine the effect of the sock to be developed with wearable technology for patients who will undergo TUR surgery on the development of hypothermia and VTE. The population of the study will consist of patients who will undergo TUR surgery between 01 October 2023 and 01 October 2024. patients will be included in the study. The study was planned as a prospective, two-arm (1:1), randomised controlled, double-blind clinical trial. The data will be collected with the "Descriptive Characteristics Form" and "Hypothermia Monitoring Form". The hypothermia follow-up form includes "Shivering Level Diagnosis Form" and "Temperature Comfort Perception Scale" The descriptive variables of the patients included in the study will be expressed as mean ± standard deviation and median (maximum-minimum), percentage and frequency. In data analysis; dependent and independent t test will be used when parametric test preconditions are met. Changes in body temperature measurements obtained after wearing socks to be developed with wearable technology, repeated measurements, analysis of variance (Repeated ANOVA) if parametric, Friedman test if non-parametric, and post-hoc test will be used in intra-group multiple comparison analyses as further analysis. Post hoc power analysis will be performed after the sample size reaches 70.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of the sock to be developed with wearable technology for patients who will undergo TUR surgery on the development of hypothermia and VTE. The population of the study will consist of patients who will undergo TUR surgery between 01October 2023 and 01 October 2024. patients will be included in the study. The study was planned as a prospective, two-arm (1:1), randomised controlled, double-blind clinical trial. The data will be collected with the "Descriptive Characteristics Form" and "Hypothermia Monitoring Form". The hypothermia follow-up form includes "Shivering Level Diagnosis Form" and "Temperature Comfort Perception Scale" .Control group: Patients will be fitted with antiembolitic socks in the ward, and the control group will be fitted with the same looking socks developed before the patient is sent to the operating theatre and will be removed one day after the operation. In the study, the same-looking socks will be applied to all patients by the same coordinator. Verbal and written permission will be obtained from the patient/relative before the study is started. The data obtained from the patients will be recorded in the "Descriptive Characteristics Form" and "Hypothermia Monitoring Form" before TUR.

Study group: In addition to the routine treatment and care practices of the operating theatre, the patients included in the study group will wear antiembolytic socks and a heater sock to be developed with wearable technology. After the patients are fitted with antiembolitic socks in the ward, the socks to be developed with wearable technology will be fitted to the study group before the patient is sent to the operating theatre and will be removed one day after the operation. The socks to be used in the research (socks with the same appearance as the heating socks developed with wearable technology) will be developed by the researchers and a patent application will be made. The socks to be developed with wearable technology in the study will be applied to all patients by the same responsible researcher. Verbal and written consent will be obtained from the patient/relative before the start of the study. The data obtained from the patients will be recorded in the "Descriptive Characteristics Form" and "Hypothermia Monitoring Form" before TUR. The "Hypothermia Monitoring Form" will be filled in when the patients' vital signs are taken into the operating room, after anaesthesia is given, at the 15th, 30th and 60th minutes of the surgical procedure, at the end of the surgical procedure, when they come to the recovery room, and when they are transferred from the recovery room to the ward.The descriptive variables of the patients included in the study will be expressed as mean ± standard deviation and median (maximum-minimum), percentage and frequency. In data analysis; dependent and independent t test will be used when parametric test preconditions are met. Changes in body temperature measurements obtained after wearing socks to be developed with wearable technology, repeated measurements, analysis of variance (Repeated ANOVA) if parametric, Friedman test if non-parametric, and post-hoc test will be used in intra-group multiple comparison analyses as further analysis. Post hoc power analysis will be performed after the sample size reaches 70.

ELIGIBILITY:
Inclusion Criteria:

* Written and verbal permission to participate in the study was obtained,
* Conscious, orientated and co-operative,
* Who speaks and understands Turkish,
* Undergoing TUR surgery,
* Not hypothermic in the preoperative period,
* No peripheral vascular disease,
* Not allergic to sock material,
* Patients without devices that send electric current into the body (pacemaker, etc.)

Exclusion Criteria:

* Written and verbal permission to participate in the research could not be obtained,
* Unconscious, disorientated and uncooperative,
* Speaking Turkish and not understanding it,
* No TUR surgery,
* Hypothermic in the pre-operative period,
* With peripheral vascular disease,
* Allergic to sock material
* Patients with devices that send electric current into the body (pacemaker, etc.)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Body temperature | Perioperative period
  Hypothermia Monitoring Form: It is a form in which the body temperature, shivering level and temperature comfort perception of the patients and the time when the body temperature reached 360C in the postoperative period are recorded. Body temperature is recorded preoperatively (when the patient comes to the operating theatre preop preparation room, when the patient is taken to the operating room), intraoperatively (when anaesthesia is given, at the 30th and 60th minutes of the surgical intervention, at the end of the surgery). The level of shivering and temperature comfort perception will be measured preoperatively (when the patient comes to the operating theatre preop preparation room, when the patient is taken to the operating room) and postoperatively (when the patient comes to the recovery room, when the patient is transferred from the recovery room to the ward).
Shivering level | Perioperative period
  Tremor Level Diagnosis Form: The form, which Badjaita et al. (2008) determined the criteria by observation, determines the level of tremor according to the tremor in the extremities between 0 (no tremor) and 3 (severe tremor in the trunk, lower and upper extremities) points.
Comfort perception | Perioperative period
  Temperature Comfort Perception Scale: It is a visual analogue scale developed by Wagner (2006) to provide objective assessment of temperature comfort perception. In the scale, the level of temperature comfort perception is evaluated between 0 (extremely cold) - 10 (extremely hot) according to the patient's report.

SECONDARY OUTCOMES:
Development of venous thromboembolism | Perioperative period
  Descriptive Characteristics Form: In the form prepared by the researchers in line with the literature, VTE development status will be questioned and recorded during hospitalisation.
Descriptive Characteristics | Perioperative period
  Descriptive Characteristics Form: The form created by the researcher in line with the literature consists of questions about the age, gender, educational status of the patients and the characteristics of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Uğraş, Assoc. Dr., Study Director — Mersin University; Evren Değirmenci, Assoc.Dr., Principal Investigator — Mersin University; Murat Bozlu, Prof. Dr., Principal Investigator — Mersin University

IPD SHARING:
Plan to Share IPD: No
All datasets will support enriched data to be available and accessible online. Aperta Turkey Open Archive is a platform where data uploads are made by researchers, called a data repository, which can be used free of charge and provides data management, protection and storage. Since publications will be obtained from these data produced during the project, it is planned to be shared in APERTA, the Open Archive of TÜBİTAK, in line with FAIR principles (findable, accessible, interoperable, reusable) and the data will be reused for new research

REFERENCES:
- [Background] Leslie SW, Chargui S, Stormont G. Transurethral Resection of the Prostate. 2023 Sep 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560884/ PMID 32809719
- [Background] Kim LHC, Patel MI. Transurethral resection of bladder tumour (TURBT). Transl Androl Urol. 2020 Dec;9(6):3056-3072. doi: 10.21037/tau.2019.09.38. PMID 33457279
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Health Statistics Yearbook. (2020). Access address: https://dosyasb.saglik.gov.tr/Eklenti/43399 ,siy2020-tur-26052022pdf.pdf?0. Access date: 28.02.2023
- [Background] Bhindi B, Kool R, Kulkarni GS, Siemens DR, Aprikian AG, Breau RH, Brimo F, Fairey A, French C, Hanna N, Izawa JI, Lacombe L, McPherson V, Rendon RA, Shayegan B, So AI, Zlotta AR, Black PC, Kassouf W. Canadian Urological Association guideline on the management of non-muscle-invasive bladder cancer - Full-text. Can Urol Assoc J. 2021 Aug;15(8):E424-E460. doi: 10.5489/cuaj.7367. No abstract available. PMID 33938798
- [Background] Lerner LB, McVary KT, Barry MJ, Bixler BR, Dahm P, Das AK, Gandhi MC, Kaplan SA, Kohler TS, Martin L, Parsons JK, Roehrborn CG, Stoffel JT, Welliver C, Wilt TJ. Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: AUA GUIDELINE PART I-Initial Work-up and Medical Management. J Urol. 2021 Oct;206(4):806-817. doi: 10.1097/JU.0000000000002183. Epub 2021 Aug 13. PMID 34384237
- [Background] Wang JW, Man LB. Transurethral resection of the prostate stricture management. Asian J Androl. 2020 Mar-Apr;22(2):140-144. doi: 10.4103/aja.aja_126_19. PMID 31898584
- [Background] Keramidas ME, Musizza B, Kounalakis SN, Mekjavic IB. Enhancement of the finger cold-induced vasodilation response with exercise training. Eur J Appl Physiol. 2010 May;109(1):133-40. doi: 10.1007/s00421-010-1374-1. Epub 2010 Feb 5. PMID 20135142
- [Background] Association of Perioperative Registered Nurses (AORN). (2018). Guideline quick vew: venous thromboembolism. AORN, 107(2), 281-285
- [Background] Chopra, A., Singhal, A., (2021). Understanding the Wearable Technology. Proceedings of the International Conference on Innovative Computing & Communication (ICICC), http://dx.doi.org/10.2139/ssrn.3833316.
- [Background] Shei RJ, Holder IG, Oumsang AS, Paris BA, Paris HL. Wearable activity trackers-advanced technology or advanced marketing? Eur J Appl Physiol. 2022 Sep;122(9):1975-1990. doi: 10.1007/s00421-022-04951-1. Epub 2022 Apr 21. PMID 35445837
- [Background] Guk K, Han G, Lim J, Jeong K, Kang T, Lim EK, Jung J. Evolution of Wearable Devices with Real-Time Disease Monitoring for Personalized Healthcare. Nanomaterials (Basel). 2019 May 29;9(6):813. doi: 10.3390/nano9060813. PMID 31146479
- [Background] Gura V, Rivara MB, Bieber S, Munshi R, Smith NC, Linke L, Kundzins J, Beizai M, Ezon C, Kessler L, Himmelfarb J. A wearable artificial kidney for patients with end-stage renal disease. JCI Insight. 2016 Jun 2;1(8):e86397. doi: 10.1172/jci.insight.86397. PMID 27398407
- [Background] Pickham D, Berte N, Pihulic M, Valdez A, Mayer B, Desai M. Effect of a wearable patient sensor on care delivery for preventing pressure injuries in acutely ill adults: A pragmatic randomized clinical trial (LS-HAPI study). Int J Nurs Stud. 2018 Apr;80:12-19. doi: 10.1016/j.ijnurstu.2017.12.012. Epub 2017 Dec 30. PMID 29331656
- [Background] Vural F, Celik B, Deveci Z, Yasak K. Investigation of inadvertent hypothermia incidence and risk factors. Turk J Surg. 2018 Dec 1;34(4):300-305. doi: 10.5152/turkjsurg.2018.3992. PMID 30664429
- [Background] Duman A, & Yilmaz E (2016). Ortopedi ameliyatlarında perioperatif hipotermi insidansı ve risk etmenleri. Çukurova Üniversitesi Tıp Fakültesi Dergisi, 41(4), 687 - 694.
- [Background] Yüksel, S. & Altun Uğraş, G. (2016). Cerrahi hastasında hipotermi gelişimini önlemede hemşirenin rolü. Mersin Üniversitesi Sağlık Bilimleri Dergisi, 9 (2), 113-121. https://dergipark.org.tr/tr/pub/mersinsbd/issue/24537/259943.
- [Background] Özsoy H. (2022). Total diz artroplastisi öncesi aktif ısıtmanın ameliyat sırası vücut sıcaklığı ve konfora etkisi (Doktora Tezi). Ege Üniversitesi Sağlık Bilimleri Enstitüsü. İzmir.
- [Background] Çam T. (2018). Kardiyovasküler cerrahi yoğun bakım hastalarında endotrakeal tüp tespitinde kullanılan yöntemlerin aspirasyon sırasındaki hemodinamik değişkenlere etkisi. (Yüksek Lisans Tezi). Mersin Üniversitesi Sağlık Bilimleri Enstitüsü. Mersin.
- [Background] Sari S, Aksoy SM, But A. The incidence of inadvertent perioperative hypothermia in patients undergoing general anesthesia and an examination of risk factors. Int J Clin Pract. 2021 Jun;75(6):e14103. doi: 10.1111/ijcp.14103. Epub 2021 Feb 28. PMID 33616248
- [Background] Yi J, Xiang Z, Deng X, Fan T, Fu R, Geng W, Guo R, He N, Li C, Li L, Li M, Li T, Tian M, Wang G, Wang L, Wang T, Wu A, Wu D, Xue X, Xu M, Yang X, Yang Z, Yuan J, Zhao Q, Zhou G, Zuo M, Pan S, Zhan L, Yao M, Huang Y. Incidence of Inadvertent Intraoperative Hypothermia and Its Risk Factors in Patients Undergoing General Anesthesia in Beijing: A Prospective Regional Survey. PLoS One. 2015 Sep 11;10(9):e0136136. doi: 10.1371/journal.pone.0136136. eCollection 2015. PMID 26360773
- [Background] Badjatia N, Strongilis E, Gordon E, Prescutti M, Fernandez L, Fernandez A, Buitrago M, Schmidt JM, Ostapkovich ND, Mayer SA. Metabolic impact of shivering during therapeutic temperature modulation: the Bedside Shivering Assessment Scale. Stroke. 2008 Dec;39(12):3242-7. doi: 10.1161/STROKEAHA.108.523654. Epub 2008 Oct 16. PMID 18927450
- [Background] Wagner D, Byrne M, Kolcaba K. Effects of comfort warming on preoperative patients. AORN J. 2006 Sep;84(3):427-48. doi: 10.1016/s0001-2092(06)63920-3. PMID 17004666